CLINICAL TRIAL: NCT00497783
Title: Safety Dermatological Evaluation of the Acceptability With Gynecological Follow up for Dermacyd Femina Delicata
Brief Title: Acceptability Lactoserum (Dermacyd Delicata - New Fragrance)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LACTO_L_02949
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2008-05-20 (Estimated); Status verified 2008-05

CONDITIONS: Hygiene
MeSH Terms: interventions — lactoserum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Lactoserum

SUMMARY:
The purpose of this study is to demonstrate the safety of the gynecological formulation in normal and usual usage condition of Dermacyd Femina Delicata.

ELIGIBILITY:
Inclusion Criteria:

* Integral skin in the tested region

Exclusion Criteria:

* Pregnancy or breastfeeding women
* Use of Anti-inflammatory or immune-suppression drugs
* Topical medication use at the tested region
* Active cutaneous gynaecological disease which may interfere in study results
* Personal history of allergic disease at the area to be treated
* Allergic or atopic history

The above information is not intended to contain considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-05

PRIMARY OUTCOMES:
Clinical and local tolerability | 21 days
Adverse events and their association with the treatment. | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Jaderson Lima, Study Director — Sanofi
Locations (1):
- Sanofi-aventis, São Paulo, Brazil